CLINICAL TRIAL: NCT03166397
Title: A Phase 2, Single-Center, Open Label Study of Autologous, Adoptive Cell Therapy Following a Reduced Intensity, Non-myeloablative, Lymphodepleting Induction Regimen in Metastatic Melanoma Patients
Brief Title: Adoptive Cell Therapy Following a Non-myeloablative, Lymphodepleting Induction Regimen in Metastatic Melanoma Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-16-3566-JS-CTIL
Record Dates: First submitted 2017-05-21; First posted 2017-05-25 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Malignant Melanoma Stage IV
MeSH Terms: conditions — Melanoma | interventions — fludarabine; Cyclophosphamide; Interleukin-2; Nivolumab; Ipilimumab; FMT protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACT TIL (Experimental): 1. Reduced Intensity, non-myeloablative, lymphodepleting induction regimen using Cyclophosphamide 30mg/kg/day with Fludarabine (25 mg/m2/d) followed by 3 consecutive days of Fludarabine 25mg/m2/d..
  2. Preparation and administration of TIL
  3. Bolus high-dose (720,000 IU/kg) IL-2 will be administered to each patient every 8 hours, to tolerance. A maximum of 10 doses will be administered per patient.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: TIL; Drug: IL-2
- ACT TIL + Anti PD-1 (Experimental): 1. Single dose of Nivolumab 480 mg fixed dose
  2. Reduced Intensity, non-myeloablative, lymphodepleting induction regimen using Cyclophosphamide 30mg/kg/day with Fludarabine (25 mg/m2/d) followed by 3 consecutive days of Fludarabine 25mg/m2/d..
  3. Preparation and administration of TIL
  4. Bolus high-dose (720,000 IU/kg) IL-2 will be administered to each patient every 8 hours, to tolerance. A maximum of 10 doses will be administered per patient.
  5. Second dose of Nivolumab 480 mg fixed dose (at least 4 weeks from the first dose)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: TIL; Drug: IL-2; Drug: Nivolumab
- ACT TIL FMT + Anti CTLA4 (Experimental): 1. FMT loading dose given via colonoscopy
  2. FMT 12 oral capsules as maintenance - given 2 times
  3. Single dose of Ipilimumab 1mg/kg up to 100 mg
  4. Reduced Intensity, non-myeloablative, lymphodepleting induction regimen using Cyclophosphamide 30mg/kg/day with Fludarabine (25 mg/m2/d) followed by 3 consecutive days of Fludarabine 25mg/m2/d..
  5. Preparation and administration of TIL
  6. Bolus high-dose (720,000 IU/kg) IL-2 will be administered to each patient every 8 hours, to tolerance. A maximum of 10 doses will be administered per patient.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: TIL; Drug: IL-2; Drug: Ipilimumab; Drug: FMT Protocol

INTERVENTIONS:
Drug: Fludarabine — Cyclophosphamide 30mg/kg/day with Fludarabine (25 mg/m2/d) followed by 3 consecutive days of Fludarabine 25mg/m2/d.
Drug: Cyclophosphamide — Cyclophosphamide 30mg/kg/day with Fludarabine (25 mg/m2/d) followed by 3 consecutive days of Fludarabine 25mg/m2/d.
Biological: TIL — TIL administration
Drug: IL-2 — Bolus high-dose (720,000 IU/kg) IL-2 will be administered to each patient every 8 hours, to tolerance. A maximum of 10 doses will be administered per patient.
Drug: Nivolumab — Nivolumab 480 mg fixed dose
  Arms: ACT TIL + Anti PD-1
Drug: Ipilimumab — Ipilimumab 1 mg/kg up to 100 mg
  Arms: ACT TIL FMT + Anti CTLA4
Drug: FMT Protocol — FMT given both directly into the colon via colonoscopy and orally using capsules (12 capsules each time).
  FMT will be taken from melanoma patients treated with Anti PD-1 who achieved a durable response of more than 12 months.
  Arms: ACT TIL FMT + Anti CTLA4

SUMMARY:
Adoptive cell therapy (ACT) with tumor-infiltrating lymphocytes (TILs) in combination with lymphodepletion and high-dose interleukin 2 (IL-2) has demonstrated reproducible objective response rates of approximately 50 percent in patients with highly advanced, refractory metastatic melanoma.

Recent developments in theTIL ACT procedure facilitate the use of a reduced-intensity, non-myeloablative, lympho-depleting preparative regimen which is expected to be both less toxic and equally efficient compared to previous regimens.

Recently patients recruited post Anti PD-1 therapy had inferior responses in comparison to the pre immune checkpoint inhibitors era. Therefore 2 new arms were added:

1. TIL-ACT with combination of 2 doses of Nivolumab fixed dose 480mg, pre and post TIL.
2. TIL-ACT with FMT given using colonoscopy once and 2 maintenance doses of 12 orally ingested capsules, concurrently with a single dose of Ipilimumab 1 mg/kg up to 100 mg.

DETAILED DESCRIPTION:
The Sponsor is developing the ex-vivo expanded autologous TIL as the Investigational Product (IP). Yet, the administration of the TIL cellular product can only be accomplished in the context of an autologous, Adoptive Cell Therapy (ACT) procedure which is composed of the following steps:

1. Reduced Intensity, non-myeloablative, lymphodepleting induction regimen using Cyclophosphamide 30mg/kg/day with Fludarabine (25 mg/m2/d) followed by 3 consecutive days of Fludarabine 25mg/m2/d.
2. Bolus high-dose (720,000 IU/kg) IL-2, which will be administered to each patient every 8 hours, to tolerance. A maximum of 10 doses will be administered per patient.
3. Early-stage follow-up until 30 days post-discharge
4. Late-stage follow-up, such as CT scans, will be carried out four and twelve weeks after TIL administration, and then every 3 months thereafter for the first year after TIL therapy; for the second year and onwards, as clinically indicated.

Recently 2 new arms were, using the same protocol described above with the following additions:

Arm 2 - TIL-ACT + Anti PD-1 -the addition of 2 doses of Nivolumab fixed dose 480mg, pre and post TIL.

Arm 3 - TIL-ACT with FMT + Anti CTLA4 - the addition of FMT given using colonoscopy once and 2 maintenance doses of 12 orally ingested capsules, concurrently with a single dose of Ipilimumab 1 mg/kg up to 100 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Measurable metastatic Melanoma with at least one lesion that is resectable for TIL generation.
2. Refractory to standard treatment
3. Patients with one or more brain metastases less than 1 cm each, and any patients with 1 or 2 brain metastases greater than 1 cm must have been treated and stable for 6 weeks.
4. Greater than or equal to 18 years of age.
5. Willing to practice birth control from the start of chemotherapy until 120 days after release from the hospital.
6. Clinical performance status of ECOG 0 or 1
7. Hematology:

   Absolute neutrophil count greater than 1000/mm3 without support of filgrastim Normal WBC (greater than 3000/mm3). Hemoglobin greater than 8.0 g/dL Platelet count greater than 100,000/mm3
8. Serology:

   Seronegative for HIV antibody. Seronegative for Hepatitis B or Hepatitis C.
9. Chemistry:

   Serum ALT/AST less than three times the upper limit of normal (ULN). Serum creatinine less than or equal to 1.6 mg/dL Total bilirubin no more than 1.5 times the ULN, except in patients with Gilbert Syndrome who must have a total bilirubin less than 3 mg/dL.
10. Negative pregnancy test in women of child bearing potential because of the potentially dangerous effects of the preparative chemotherapy on the fetus.
11. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo). Patients may have undergone minor surgical procedures with the past 3 weeks, as long as all toxicities have recovered to grade 1 or less.

Exclusion Criteria:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the non-myeloablative, lymphodepleting induction regimen on the fetus or infant.
2. Systemic steroid therapy required.
3. Active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
4. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease and AIDS).
5. Opportunistic infections (the experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study , including history of an anaphylactic reaction to penicillin or gentamicin
7. History of coronary revascularization or ischemic symptoms
8. Any patient known to have an LVEF less than or equal to 50 percent .
9. Documented LVEF of less than or equal to 50 percent tested in patients with clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
10. Documented FEV1 and DLCO (relative to predicted) less than or equal to 60 percent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06-05 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective tumor responses | 3 years
  Radiological follow up via CT to determine the sum of Complete Responders (CR) + Partial Responders (PR) + Stable Disease (SD) as assessed by RECIST 1.1
Assess adverse events using NCI CTCAE v4.03 during treatment and follow-up | 3 years
  Adverse events will be assessed using NCI CTCAE v4.03 during treatment and follow-up

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  Overall survival is defined as the time from study entry until death from any cause
Response Rate (RR) | 3 years
  Radiological follow up via CT to determine the sum of Complete Responders (CR) + Partial Responders (PR) as assessed by RECIST 1.1
Progression-Free Survival (PFS) | 3 years
  Progression free survival according to RECIST 1.1
Quality of Life (QoL) | 3 years
  Assessment of QoL using the EORTC QLQ-MEL38 instrument (specific for Melanoma)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided
To be considered

REFERENCES:
- [Derived] Nissani A, Lev-Ari S, Meirson T, Jacoby E, Asher N, Ben-Betzalel G, Itzhaki O, Shapira-Frommer R, Schachter J, Markel G, Besser MJ. Comparison of non-myeloablative lymphodepleting preconditioning regimens in patients undergoing adoptive T cell therapy. J Immunother Cancer. 2021 May;9(5):e001743. doi: 10.1136/jitc-2020-001743. PMID 33990415